CLINICAL TRIAL: NCT05159518
Title: A Phase 1, Open-Label, Multicenter, Dose Escalation and Confirmation Study of PRT2527 in Participants With Advanced Solid Tumors
Brief Title: A Study of PRT2527 in Participants With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prelude Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRT2527-01
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Sarcoma; Castrate Resistant Prostate Cancer; Hormone Receptor Positive HER2 Negative Breast Cancer; Non-small Cell Lung Cancer; Solid Tumors With Known MYC Amplification
Keywords: Breast Cancer; Castrate Resistant Prostate Cancer; CDK9 Inhibitor; CRPC; Cyclin-dependent Kinase 9; Hormone Receptor Positive HER2 Negative Breast Cancer; HR+/HER2- Breast Cancer; Non-small Cell Lung Cancer; NSCLC; Prostate Cancer; PRT2527; Refractory Solid Tumors; Relapsed Solid Tumors; Sarcoma
MeSH Terms: conditions — Sarcoma; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRT2527 (Experimental): PRT2527 will be administered by intravenous infusion
  Interventions: Drug: PRT2527

INTERVENTIONS:
Drug: PRT2527 — PRT2527 will be administered by intravenous infusion

SUMMARY:
This is a Phase 1 dose-escalation and confirmation study of PRT2527, a Cyclin-dependent Kinase 9 (CDK9) inhibitor, in participants with advanced solid tumors. The purpose of this study is to define the dosing schedule, and maximally tolerated dose to be used in subsequent development of PRT2527.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalation and confirmation Phase 1 study of PRT2527, a CDK9 inhibitor, evaluating participants with selected advanced/metastatic sarcomas displaying a documented gene fusion, castrate resistant prostate cancer, hormone receptor positive HER2-negative breast cancer, advanced/metastatic non-small cell lung cancer, and solid tumors displaying MYC amplification. The study plan expects to evaluate approximately six dose levels of approximately 1-6 participants per dose level; however additional and/or intermediate dose levels may be explored. Taking into account pharmacokinetic and pharmacodynamic data from the preceding dose levels, the dose may be escalated until a dose limiting toxicity is identified. The total sample size will be approximately 30 patients for MTD and RP2D determination.

ELIGIBILITY:
Inclusion Criteria:

* Tumor types under study

  1. Selected sarcomas with a documented gene fusion
  2. Castrate resistant prostate cancer (CRPC)
  3. Hormone receptor positive (HR+), HER2 negative (HER2-) breast cancer
  4. Non-small cell lung cancer (NSCLC)
  5. MYC amplified solid tumors
* Must have measurable disease per RECIST 1.1; participants with CRPC or sarcoma may have nonmeasurable but evaluable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1
* Adequate organ function
* Must provide tumor tissue sample to the central laboratory for biomarker analysis
* Participants must have recovered from the effects of prior cancer-related therapy, radiotherapy, or surgery to ≤ Grade 1

Exclusion Criteria:

* Primary malignancies of the CNS, or uncontrolled CNS metastases, including impending spinal cord compression
* have a corrected QT interval >480 msec from prior or baseline
* have impaired cardiac function or clinically significant cardiac disease
* Treatment with strong inhibitors or inducers of CYP3A4
* Prior exposure to a CDK9 inhibitor
* History of another malignancy except for:

  1. Curatively treated malignancy with no known active disease
  2. Curatively treated non-melanoma skin cancer without evidence of disease
  3. Curatively treated carcinoma in situ without evidence of disease
* have undergone major surgery within 2 weeks prior to Week 1 Day 1
* have had chemotherapy, biologic therapy, targeted therapy, immunotherapy, extended-field radiotherapy, or investigational agents within 5 half-lives or 28 days (whichever is shorter) prior to administration of the first dose of study drug on Week 1 Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) of PRT2527 | Baseline through Day 21
  Dose limiting toxicities will be evaluated over the 21-day observation period
Maximally tolerated dose (MTD) of PRT2527 | Baseline through approximately 1 year
  The MTD will be established for further investigation in participants with advanced solid tumors
Recommended phase 2 dose (RP2D) and schedule of PRT2527 | Baseline through approximately 1 year
  The RP2D will be established for further investigation in participants with advanced solid tumors

SECONDARY OUTCOMES:
Safety and tolerability of PRT2527: AEs, SAEs, CTCAE assessments | Baseline through approximately 2 years
  Safety and tolerability will be assessed by recording adverse events (AEs) and serious adverse events (SAEs) according to Common Terminology Criteria for Adverse Events (CTCAE)
Pharmacokinetic profile of PRT2527: maximum observed plasma concentration | Baseline through approximately 1 year
  PRT2527 pharmacokinetics will be calculated including the maximum observed plasma concentration
Anti-tumor activity of PRT2527: measurement of objective responses | Baseline through approximately 2 years
  Anti-tumor activity of PRT2527 based on the measurement of objective responses to PRT2527 according to the disease-specific response criteria for patients with advanced solid tumors
Duration of response to PRT2527: Objective responses | Baseline through approximately 2 years
  Duration of response will be calculated for all patients eligible for response determination from the time that a response is first observed until progression or death, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Investigational Drug Services, AdventHealth Celebration, Celebration, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mary Crowley Cancer Research, Dallas, Texas
  - NEXT Virginia, Fairfax, Virginia